CLINICAL TRIAL: NCT01395017
Title: Placebo-controlled Double-blind Trial of Dasatinib Added to Gemcitabine for Subjects With Locally-advanced Pancreatic Cancer
Brief Title: Dasatinib Added to Gemcitabine for Subjects With Locally-advanced Pancreatic Cancer
Acronym: LAPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 287-11-201
Record Dates: First submitted 2011-07-08; First posted 2011-07-15 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Dasatinib; chemotherapy; Locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): One arm will receive standard of care treatment (ie, GEM 1000 mg/m2 by intravenous [IV] infusion weekly for 3 weeks of a 4-week cycle) plus dasatinib 100 mg by mouth once daily (QD).
  Interventions: Drug: dasatinib
- Group 2 (Placebo Comparator): The other arm will receive standard of care treatment (ie, GEM 1000 mg/m2 by intravenous [IV] infusion weekly for 3 weeks of a 4-week cycle) plus matched placebo by mouth once daily (QD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dasatinib — GEM 1000 mg/m2 by intravenous [IV] infusion weekly for 3 weeks of a 4-week cycle plus dasatinib 100 mg (or matched placebo) by mouth once daily (QD). Subjects will continue to receive study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: BMS-354825
  Arms: Group 1
Drug: Placebo — Matching Placebo
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine whether patients with locally advanced pancreatic cancer who receive dasatinib added to standard of care (gemcitabine) live longer, compared to patients who receive standard of care (gemcitabine) plus placebo; i.e. gemcitabine alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic documentation of unresectable adenocarcinoma of the pancreas.
* Recovery from toxicity of previous procedures to establish the diagnosis. ECOG PS 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Evidence of metastatic disease.
* Previous radiotherapy or chemoradiotherapy.
* History of or current pleural effusion.
* History of significant cardiovascular disease.
* Clinically significant bleeding disorder or coagulopathy.
* Concomitant medication with strong CYP 3A4 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (11):
  - Birmingham, Alabama
  - Los Angeles, California
  - Orange, California
  - San Francisco, California
  - Aurora, Colorado
  - Boynton Beach, Florida
  - Tampa, Florida
  - Wichita, Kansas
  - Minneapolis, Minnesota
  - Albuquerque, New Mexico
  - Bethlehem, Pennsylvania
- Australia (6):
  - Blacktown, New South Wales
  - Liverpool, New South Wales
  - Tweed Heads, New South Wales
  - Footscray, Victoria
  - Frankston, Victoria
  - Parkville, Victoria
- Vienna, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (4):
  - Olomouc
  - Pardubice
  - Prague
  - Zlín
- France (9):
  - Clermont-Ferrand, Auvergne
  - Paris, Cedex 14
  - Angers, Maine-et-Loire
  - Saint-Priest-en-Jarez, Pays de la Loire Region
  - Besançon
  - Clichy
  - Lille
  - Lyon
  - Saint-Priest-en-Jarez
- Germany (4):
  - Tübingen, Baden-Wurttemberg
  - Cologne
  - Hamburg
  - München
- Hungary (3):
  - Pécs, Baranya
  - Budapest
  - Győr
- Dublin, Ireland
- Italy (4):
  - Milan, MI
  - Udine, UD
  - Ancona
  - Reggio Emilia
- Poland (3):
  - Jelenia Góra
  - Lublin
  - Olsztyn
- Romania (3):
  - Bucharest, Bucharest
  - Craiova, Dolj
  - Cluj-Napoca
- Russia (5):
  - Kazan', Tatarstan Republic
  - Chelyabinsk
  - Krasnodar
  - Moscow
  - Voronezh
- United Kingdom (12):
  - Hull, East Yorks
  - Chelmsford, Essex
  - Maidstone, Kent
  - Northwood, Middlesex
  - Sutton, Surrey
  - Leeds, West Yorkshire
  - Edinburgh
  - Glasgow
  - Liverpool
  - London
  - Metropolitan Borough of Wirral
  - Salisbury

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 202 participants were enrolled at 79 study sites in 15 countries.
Pre-assignment Details: Participants were randomly assigned in a 1:1 ratio to receive dasatinib + gemcitabine (GEM) or placebo + GEM. Participants were stratified at the time of randomization by baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (0 versus 1) and intent to receive radiotherapy (RT) (yes or no).
Groups:
- Dasatinib + GEM: GEM 1000 mg/m2 by intravenous (IV) infusion weekly for 3 weeks of a 4-week cycle plus dasatinib 100 mg by mouth once daily (QD).
- Placebo + GEM: GEM 1000 mg/m2 by IV infusion weekly for 3 weeks of a 4-week cycle plus matched placebo by mouth QD.
Period: Overall Study
Arm/Group | Dasatinib + GEM | Placebo + GEM
Started | 100 | 102
Treated | 98 | 101
Completed | 0 | 0
Not Completed | 100 | 102
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 26 | 12
Not completed — Physician Decision | 11 | 15
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Protocol deviation | 1 | 2
Not completed — Death | 4 | 3
Not completed — Disease progression | 42 | 58
Not completed — Sponsor discontinued study | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib + GEM: GEM 1000 mg/m2 by IV infusion weekly for 3 weeks of a 4-week cycle plus dasatinib 100 mg by mouth QD.
- Total: Total of all reporting groups
Arm/Group | Dasatinib + GEM | Placebo + GEM | Total
Number analyzed (Participants) | 100 | 102 | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (9.1) | 64.7 (9.6) | 64.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 56 | 99
  Male | 57 | 46 | 103

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) is the time from randomization until time of death from any cause by 02 December 2013.
Time Frame: From randomization until date of death from any cause by 02 December 2013
Population: The intent-to-treat (ITT) data which was composed of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dasatinib + GEM | Placebo + GEM
Number analyzed (Participants) | 100 | 102
Days | 375 [310 to 450] | 393 [356 to 467]
Statistical Analysis 1: Comparison: Dasatinib + GEM vs Placebo + GEM; Using a 1-sided alpha=0.2, a population of 200 participants (100 GEM plus dasatinib and 100 GEM plus placebo) has 79% power to show an increase in median OS from 10 to 13.3 months (hazard ratio [HR] =0.75, assuming analysis of 135 deaths); Test type: Superiority or Other; p = 0.3864, Cox proportional hazard model — The log-rank test was used to test OS. As a sensitivity analysis, HR and its confidence interval was also provided for OS using the Cox proportional hazard model; Adjusting for baseline factors - treatment, ECOG PS, region, CA19-9 level (< 1000 IU/mL or >/=1000 IU/mL), and RT during trial (yes or no); Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.85 to 1.65]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS - time from randomization to unequivocal local or distant disease progression, death or discontinuation from trial for any reason by 02 December 2013. Progression events were determined according to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 every 8 weeks.
Time Frame: Time from randomization to earliest PFS event by 02 December 2013
Population: The ITT data which was composed of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dasatinib + GEM | Placebo + GEM
Number analyzed (Participants) | 100 | 102
Days | 167 [114 to 212] | 166 [160 to 199]
Statistical Analysis 1: Comparison: Dasatinib + GEM vs Placebo + GEM; Trial has 88% power to show a median PFS increase from 5 to 7 months (with 1-sided alpha=0.15, total 176 events, HR=0.714); Test type: Superiority or Other; p = 0.6761, Cox proportional hazard model — The log-rank test was used to test PFS. As a sensitivity analysis, HR and its confidence interval was also provided for PFS using the Cox proportional hazard model; Adjusting for baseline factors: treatment, ECOG PS, region, CA19-9 level (< 1000 IU/mL or >/=1000 IU/mL), and RT during trial (yes or no); Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.73 to 1.34]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from randomization, throughout each treatment cycle to final study visit. Follow-up visits conducted until all ongoing AEs resolved or clinically stable.
Description: The safety data set (participants who received at least one dose of study treatment) included 98 participants in the Dasatinib + GEM group and 101 participants in the placebo + GEM group.
Arm/Group | Dasatinib + GEM | Placebo + GEM
Serious Adverse Events (participants affected / at risk) | 53/98 | 48/101
Other Adverse Events (participants affected / at risk) | 93/98 | 98/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib + GEM (N=98) | Placebo + GEM (N=101)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 3 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Small intestine obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 0 | 1
Device occlusion (General disorders) | 5 | 5
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 4
Stent malfunction (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 4 | 2
Bile duct stenosis (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 4 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Liver abcess (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Necrolytic migratory erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib + GEM (N=98) | Placebo + GEM (N=101)
Anemia (Blood and lymphatic system disorders) | 50 | 28
Leukopenia (Blood and lymphatic system disorders) | 8 | 13
Lymphopenia (Blood and lymphatic system disorders) | 5 | 7
Neutropenia (Blood and lymphatic system disorders) | 53 | 49
Thrombocytopenia (Blood and lymphatic system disorders) | 38 | 39
Abdominal pain (Gastrointestinal disorders) | 33 | 36
Abdominal pain upper (Gastrointestinal disorders) | 10 | 18
Ascites (Gastrointestinal disorders) | 8 | 6
Constipation (Gastrointestinal disorders) | 33 | 28
Diarrhoea (Gastrointestinal disorders) | 41 | 29
Dry mouth (Gastrointestinal disorders) | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 9 | 7
Flatulence (Gastrointestinal disorders) | 6 | 11
Nausea (Gastrointestinal disorders) | 65 | 49
Stomatitis (Gastrointestinal disorders) | 9 | 8
Vomiting (Gastrointestinal disorders) | 40 | 34
Asthenia (General disorders) | 17 | 16
Chest pain (General disorders) | 2 | 7
Chills (General disorders) | 6 | 4
Face oedema (General disorders) | 5 | 1
Fatigue (General disorders) | 50 | 46
Oedema peripheral (General disorders) | 32 | 22
Pain (General disorders) | 2 | 8
Pyrexia (General disorders) | 22 | 27
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 7
Nasopharyngitis (Infections and infestations) | 7 | 5
Oral candidiasis (Infections and infestations) | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 3
Urinary tract infection (Infections and infestations) | 6 | 1
Alanine aminotransferase increased (Investigations) | 22 | 14
Aspartate aminotransferase increased (Investigations) | 16 | 11
Blood alkalne phosphatase increased (Investigations) | 15 | 8
Blood bilirubin increased (Investigations) | 13 | 6
Gamma glutamyltransferase increased (Investigations) | 5 | 1
Haemaglobin decreased (Investigations) | 5 | 6
Neutrophil count decreased (Investigations) | 6 | 5
Platelet count decreased (Investigations) | 7 | 4
Weight decreased (Investigations) | 21 | 11
White blood cell count decreased (Investigations) | 8 | 2
Decreased appetite (Metabolism and nutrition disorders) | 48 | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 16
Muscloskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 5
Dizziness (Nervous system disorders) | 4 | 11
Dysgeusia (Nervous system disorders) | 12 | 6
Headache (Nervous system disorders) | 12 | 9
Anxiety (Psychiatric disorders) | 10 | 4
Depression (Psychiatric disorders) | 6 | 5
Insomnia (Psychiatric disorders) | 12 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 19
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 20 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 9
Rash (Skin and subcutaneous tissue disorders) | 20 | 14
Hypertension (Vascular disorders) | 4 | 10

LIMITATIONS AND CAVEATS:
5 participants (who had not experienced disease progression at the time of event-driven data cut-off) were told the study results and were instructed to indicate "sponsor discontinued study" if they did not want to continue in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No